CLINICAL TRIAL: NCT03840096
Title: Effect of Augmenting a Standard Total Knee Pathway Protocol With a 12-week Peri-Operative Program of BREG Flex
Brief Title: Effectiveness of BREG Flex in 12-week Peri-operative Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hawkins Foundation (Other)
Collaborators: BREG, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00075229
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Quadriceps NMES using Breg Flex (Experimental)
  Interventions: Device: Breg Flex
- Control (No Intervention)

INTERVENTIONS:
Device: Breg Flex — All subjects in the treatment group will receive quadriceps Neuro Muscular Electrical Stimulation using Breg Flex device on the affected leg to guide and monitor of knee HEP during the 6 weeks prior to surgery and 12 weeks following surgery.
  Arms: Quadriceps NMES using Breg Flex

SUMMARY:
Patient outcomes following total knee replacement and standard physical therapy will be compared between subjects who use the Breg Flex study device vs those who do not. Subjects will be evaluated for knee range of motion, strength and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are scheduled for Total Knee Arthroplasty by a single surgeon (Burnikel)
2. Individuals who are at least 55 years of age
3. Individuals with a body mass index (BMI) <45
4. Must be able and willing to complete all study assessments and to be followed for the full course of the study.
5. Must be able to read, write and follow instructions in English.
6. Must be able and willing to provide informed consent.
7. Must be willing and able to attend the pre-op assessment

Exclusion Criteria:

1. Individuals with a history of any underlying neurological conditions
2. Individuals with a history of stroke
3. Individuals with a history of neurological disorder that affects lower extremity function (stroke, peripheral neuropathy, Parkinson's disease, multiple sclerosis, etc.)
4. Individuals with physical conditions which would make them unable to perform study procedures
5. Pregnant women or inadequate precautions to prevent pregnancy
6. Diagnosis of a medical condition that would contraindicate treatment with the product, e.g. skin lesions at electrode site.
7. Individuals with a diagnosis of inflammatory arthritis (Rheumatoid arthritis, gout or psoriatic arthritis)?
8. Individuals with muscle diseases (i.e. muscular dystrophy)
9. Visible skin injury or disease on their legs
10. Principal investigator for this study, or member of study staff

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Patient Acceptable Symptoms State (PASS) | 52 weeks post op
  Patient reported outcome recording patient satisfaction with level of recovery. Patients report that they are either satisfied or not.

SECONDARY OUTCOMES:
Knee Osteoarthritis Outcome Score-JR (KOOS-JR) | 6 week and 1 week preoperatively and 3 ,6, 12, 52 week post op
  Patient reported outcome measuring knee joint specific pain and physical function. The answer values range from none to extreme to describe pain and physical limitation.
Number of Participant Physical Therapy Visits | 3 ,6, 12, 52 week post op
  The number of Physical therapy visits between data collection time points
Range of motion | 6 week and 1 week preoperatively and 3 ,6, 12 week post op
  Passive flexion and extension range of motion of knee
Strength | 6 week and 1 week preoperatively and 3 ,6, 12 week post op
  Strength of quadriceps as measured on Biodex

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - ATI Physical Therapy, Greenville, South Carolina
  - Steadman Hawkins Clinic of the Carolinas - Greenville Health System, Greenville, South Carolina